CLINICAL TRIAL: NCT02743949
Title: A Randomized, Double-Blind, Proof-of-Concept, Phase 2 Study to Evaluate the Efficacy and Safety of Once Daily Oral Vonoprazan 20 mg or Vonoprazan 40 mg Compared to Esomeprazole 40 mg for the Treatment of Subjects With Symptomatic Gastro-Esophageal Reflux Disease Who Have a Partial Response Following Treatment With a High Dose of Proton Pump Inhibitor
Brief Title: Comparison of Vonoprazan to Esomeprazole in Participants With Symptomatic GERD Who Responded Partially to a High Dose of Proton Pump Inhibitor (PPI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vonoprazan-2001; U1111-1172-2373 (Registry Identifier: WHO); 2015-001154-14 (EudraCT Number); 16/LO/0285 (Registry Identifier: NRES)
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Gastroesophageal Reflux
Keywords: Drug therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esomeprazole 40 mg (Active Comparator): Esomeprazole 40 mg over-encapsulated tablets, orally, once daily for 4 weeks then esomeprazole placebo-matching capsules, orally, once daily for 2 weeks during the run-in period, followed by esomeprazole 40 mg, over encapsulated tablets, orally, once daily for 4 weeks during the active treatment period.
  Interventions: Drug: Vonoprazan; Drug: Esomeprazole; Drug: Esomeprazole Placebo
- Vonoprazan 20 mg (Experimental): Esomeprazole 40 mg over-encapsulated tablets, orally, once daily for 4 weeks then esomeprazole placebo-matching capsules, orally, once daily for 2 weeks during the run-in period, followed by vonoprazan 20 mg, over-encapsulated capsules, orally, once daily for 4 weeks during the treatment period.
  Interventions: Drug: Vonoprazan; Drug: Esomeprazole; Drug: Esomeprazole Placebo
- Vonoprazan 40 mg (Experimental): Esomeprazole 40 mg over-encapsulated tablets, orally, once daily for 4 weeks then esomeprazole placebo-matching capsules, orally, once daily for 2 weeks during the run-in period, followed by vonoprazan 40 mg, over-encapsulated capsules, orally, once daily for 4 weeks during the active treatment period.
  Interventions: Drug: Esomeprazole; Drug: Esomeprazole Placebo

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan over-encapsulated capsules
  Other Names: TAK-438
  Arms: Esomeprazole 40 mg; Vonoprazan 20 mg
Drug: Esomeprazole — Esomeprazole over-encapsulated tablets
Drug: Esomeprazole Placebo — Esomeprazole placebo-matching capsules

SUMMARY:
The purpose of this study is to determine the effect of vonoprazan compared to esomeprazole for preventing heartburn symptoms over a 4-week treatment period in participants who have a partial response to treatment with esomeprazole.

DETAILED DESCRIPTION:
The drug being tested in this study is called vonoprazan. Vonoprazan is being tested to treat people who have symptomatic gastroesophageal reflux disease (GERD) with a partial response to treatment with a high dose of esomeprazole. This study will look at improvement in heartburn symptoms in participants who take vonoprazan compared to esomeprazole.

The study will enroll approximately 213 patients. All participants will receive esomeprazole or esomeprazole placebo-matching capsules (this is a capsule that looks like esomeprazole but has no active ingredient) during a 7-week run-in period. Participants will then be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Esomeprazole 40 mg
* Vonoprazan 20 mg
* Vonoprazan 40 mg

All participants will be asked to take one capsule at the same time each day throughout the study. All participants will be asked to record heartburn symptoms in a diary every morning upon waking and every evening before going to sleep.

This multi-center trial will be conducted in Europe. The overall time to participate in this study is 12 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 1 week after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a man or a woman and ≥18 years of age, at the time of the Screening visit.
4. Has a documented history of symptoms of both heartburn (burning pain) and acid regurgitation prior to entry into the study.
5. The subject has a medical history of ≥ 8 weeks of persistent heartburn symptoms in the presence of regurgitation symptoms (persistent heartburn symptoms defined as heartburn symptoms on ≥ 2 days a week) that are troublesome despite appropriate and correctly performed treatment with a PPI at standard doses.
6. Is ≥85% compliant at taking their Run-in medication and completing their e-Diary. Compliance for taking the Run-in medication is defined as the medication provided (esomeprazole and placebo) taken for 85% of the 6 weeks Run-in Period (or on 36 of 42 days of the Run-in Period).Compliance for the e-Diary is defined as the percentage of scheduled assessments that are completed based on 2 assessments per day (daytime and nighttime). For randomization, 85% compliance is required and is defined as 12 of 14 assessments completed over the 7-day period (Day -21 to Day-14) prior to the single blind Placebo Run-in Period.
7. Has a partial response to a PPI defined as having heartburn on 2 to 5 days and regurgitation on at least one day of the last week (Week 4) of a 4 week PPI Run-In Period with esomeprazole 40 mg and an increase of at least 2 symptom days of heartburn in the last week of a 2 week Placebo Run-In Period (4 to 7 symptom days) and at least one symptom day with regurgitation compared with the last week of the PPI Run-In Period.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 4 weeks after last dose of the study medication.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the Screening Visit.
2. Has received vonoprazan in a previous clinical study.
3. Is an immediate family member, study site employee, is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling), or may have consented under duress.
4. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening.
5. Has a history of erosive esophagitis of Los Angeles (LA) Classification Grade B severity or worse prior to screening or at Screening endoscopy.
6. Has a history of or any coexisting diseases affecting the esophagus (eg, Barrett's esophagus, eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic trauma, or physiochemical trauma such as sclerotherapy to the esophagus.
7. Has "alarm features" in symptomatology, including odynophagia, severe dysphagia, bleeding, weight loss, anemia, and blood in stool, pointing to a possible malignant disease of the gastrointestinal (GI) tract. Participants displaying "alarm symptoms" in addition to the "typical" gastroesophageal reflux disease (GERD) symptoms may be included based on endoscopic exclusion of malignancy.
8. Has current or historical chest pain due to cardiac diseases (eg, within one year).
9. Has had surgical treatment for GERD (eg, cardiaplasty), dilation of an esophageal stricture (other than Schatzki ring) or gastric or duodenal surgery, except simple oversew of an ulcer or endoscopic polypectomy of benign polyps.
10. Has active gastric or duodenal ulcers which have been confirmed by endoscopy within 30 days prior to Screening. Gastric or duodenal erosions are not exclusionary, unless considered severe and symptomatic by the investigator.
11. Has had an acute upper gastrointestinal hemorrhage within 30 days prior to Screening.
12. Has current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition.
13. Has current or historical evidence of eosinophilic esophagitis (evidence may be based on the following: missing response to acid suppressive therapy, the presence of eosinophilia in histological probes of the esophageal mucosa, a normal pH profile of the distal esophagus, symptoms of dysphagia and food impaction). The exclusion of participants based on a predominance of the "typical" eosinophilic esophagitis symptoms only (as above) is considered acceptable. However, in participants with a predominance of "typical" symptoms and co-existing significant dysphagia and food impaction, the syndrome should be excluded by endoscopy with biopsy.
14. Has a documented history (within 6 months prior to screening) of functional dyspepsia (suggested by the presence of one or more of the following symptoms: epigastric pain, postprandial fullness or early satiety), or irritable bowel syndrome or other gastrointestinal diseases which are not acid-related, and therefore, are nonresponsive to gastric acid-blocking treatment.
15. Has a documented history of familial adenomatous polyposis.
16. Has known intolerance, hypersensitivity or allergies to any PPI or their components (including lansoprazole, dexlansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole), any component of vonoprazan, or antacid(s) selected as rescue medication for this study.
17. Has a history of alcohol abuse, illegal drug use, or drug addiction within the 12 months prior to Screening, or regularly consumes >21 units of alcohol (1 unit = 12 oz/300 mL beer, 1.5 oz/25 mL hard liquor/spirits, or 5 oz/100 mL wine) per week. Participants must have a negative drug screen at Screening.
18. Has evidence of a serious uncontrolled concomitant disease including: clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, systemic, or endocrine disease or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
19. Has planned, or is likely to require, in-patient surgery during the course of the study.
20. Has a history of cancer (except basal cell carcinoma of the skin) within 3 years prior to Screening.
21. Is known to have acquired immunodeficiency syndrome or chronic hepatitis due to any etiology.
22. Has abnormal laboratory values at Screening that suggest a clinically significant underlying disease or condition that may prevent the participant from completing the study.
23. Has an alanine aminotransferase (ALT), aspartate aminotransferase (AST) or T-bilirubin level which exceeds upper limit of normal (ULN) set by the testing laboratory at the Screening.
24. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
25. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study.
26. In the opinion of the investigator, is unable to comply with the requirements of the study or is unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (39):
- Belgium (5):
  - Medif, Gozée
  - SPRL Dr Yvan CALOZET, Grigomont
  - UZ Leuven, Leuven
  - SPRL MG Balthazar & Ballard, Natoye
  - Mortelmans, Jaak, Oostham
- Bulgaria (11):
  - DCC 'Sv. Pantaleymon' OOD, Pleven
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - NMTH "Tsar Boris III", Sofia
  - "City Clinic UMHAC" EOOD, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
- Okresni nemocniceStrakonice, Strakonice, Czechia
- Estonia (6):
  - OU Innomedica, Tallinn
  - Merekivi Perearstid OU, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Poland (11):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - NZOZ Inter-Med, Częstochowa
  - Centrum Medyczne Plejady, Krakow
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Centrum Medyczne Medyk, Rzeszów
  - Specjalistyczna Praktyka Lekarska Dr med. Marek Horynski, Sopot
  - SONOMED Sp.z o.o, Szczecin
  - Niepubliczny Zaklad Opieki Zdrowotnej Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych z, Torun
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - EMC Instytut Medyczny S.A., Wroclaw
- United Kingdom (5):
  - Plympton Health Centre, Plymouth, Devon
  - Whipps Cross University Hospital, London, Greater London
  - Sheepcot Medical Centre, Watford, Hertfordshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - CPS Research, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 33 investigative sites in Belgium, Bulgaria, Czech Republic, Estonia, Poland and United Kingdom from 14 July 2016 to 12 October 2018.
Pre-assignment Details: Participants with a symptomatic gastro-esophageal reflux disease who have a partial response following treatment with a high dose of proton pump inhibitor were enrolled in a 1:1:1 ratio to receive esomeprazole 40 mg, vonoprazan 20 mg, or vonoprazan 40 mg.
Groups:
- Esomeprazole 40 mg: Esomeprazole 40 mg over-encapsulated tablets, orally, once daily for 4 weeks then esomeprazole placebo-matching capsules, orally, once daily for 2 weeks during the run-in period, followed by esomeprazole 40 mg, over-encapsulated tablets, orally, once daily for 4 weeks during the active treatment period.
Period: Overall Study
Arm/Group | Esomeprazole 40 mg | Vonoprazan 20 mg | Vonoprazan 40 mg
Started | 86 | 85 | 85
Completed | 82 | 84 | 82
Not Completed | 4 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Significant Protocol Deviation | 2 | 0 | 1
Not completed — Voluntary Withdrawal | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized into the study, regardless of whether they received any dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 40 mg | Vonoprazan 20 mg | Vonoprazan 40 mg | Total
Number analyzed (Participants) | 86 | 85 | 85 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.94) | 52.0 (14.67) | 51.8 (14.09) | 52.6 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 51 | 152
  Male | 38 | 32 | 34 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 86 | 84 | 83 | 253
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 1 | 0 | 1
  Bulgaria | 61 | 55 | 61 | 177
  Czech Republic | 14 | 16 | 10 | 40
  Estonia | 2 | 5 | 4 | 11
  Poland | 8 | 7 | 7 | 22
  United Kingdom | 1 | 1 | 3 | 5
Smoking Status [Count of Participants; unit: Participants]
  Participant has never smoked | 50 | 53 | 53 | 156
  Participant is a current smoker | 21 | 23 | 22 | 66
  Participant is an ex-smoker | 15 | 9 | 10 | 34
Alcohol Classification [Count of Participants; unit: Participants]
  Participant has never drunk | 57 | 49 | 54 | 160
  Participant is a current drinker | 27 | 33 | 30 | 90
  Participant is an ex-drinker | 2 | 3 | 1 | 6
Alcohol Use [Count of Participants; unit: Participants]
  Less than 21 units of alcohol per week | 27 | 33 | 30 | 90
  Missing | 59 | 52 | 55 | 166
Caffeine Consumption [Count of Participants; unit: Participants]
  Yes | 60 | 67 | 68 | 195
  No | 26 | 18 | 17 | 61
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 169.9 (9.17) | 168.5 (9.07) | 168.1 (7.81) | 168.9 (8.71)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 78.78 (17.003) | 77.46 (16.353) | 75.81 (16.126) | 77.36 (16.481)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg per square meter (kg/m^2)] — Body Mass Index=weight (kg)/[height (m)^2]
  kg per square meter (kg/m^2) | 27.13 (4.611) | 27.21 (4.854) | 26.76 (5.076) | 27.03 (4.835)
Hospital Anxiety and Depression Scale (HADS) Anxiety Total [Mean (Standard Deviation); unit: score on scale] — HADS-A and HADS-D are 7-item subscales that measure the presence and severity of anxiety and depression symptoms, respectively, on a scale of 0 to 3. Total scores ≤ 7: no clinically relevant symptoms; 8 - 10: mild symptoms; 11 - 14: moderate symptoms; and ≥15 (maximum 21): more severe symptoms. Population: Data are reported for evaluable participants.
  score on scale
    number analyzed (Participants) | 85 | 84 | 85 | 254
    (all) | 6.5 (3.81) | 6.2 (3.38) | 7.0 (3.78) | 6.6 (3.67)
Depression Total [Mean (Standard Deviation); unit: score on scale] — HADS-A and HADS-D are 7-item subscales that measure the presence and severity of anxiety and depression symptoms, respectively, on a scale of 0 to 3. Total scores ≤ 7: no clinically relevant symptoms; 8 - 10: mild symptoms; 11 - 14: moderate symptoms; and ≥15 (maximum 21): more severe symptoms. Population: Data are reported for evaluable participants.
  score on scale
    number analyzed (Participants) | 85 | 84 | 85 | 254
    (all) | 5.9 (3.62) | 6.0 (3.50) | 6.2 (3.99) | 6.0 (3.70)
Is Erosive Esophagitis Present? [Count of Participants; unit: Participants]
  Yes | 30 | 28 | 17 | 75
  No | 56 | 57 | 68 | 181
If Yes, Grade of Erosive Esophagitis [Count of Participants; unit: Participants] — Per LA (Los Angeles) Classification - Grade 0: no mucosal breaks; Grade A: >/=1 mucosal breaks </=5 mm, none of which extends between the tops of the mucosal folds; Grade B: >/=1 mucosal breaks >5 mm, none of which extends between the tops of two mucosal folds; Grade C: mucosal breaks that extend between the tops of two or more mucosal folds, but which involve <75% of esophageal circumference; Grade D: mucosal breaks which involve >/=75% of esophageal circumference. Population: Participants with erosive esophagitis were graded.
  Participants
    Grade 0: number analyzed (Participants) | 30 | 28 | 17 | 75
    Grade 0 | 0 | 1 | 1 | 2
    Grade A: number analyzed (Participants) | 30 | 28 | 17 | 75
    Grade A | 30 | 27 | 16 | 73
Did the Endoscopist Visualize Findings Suggestive of Eosinophilic Esophagitis? [Count of Participants; unit: Participants]
  No | 86 | 85 | 85 | 256
H Pylori Status [Count of Participants; unit: Participants]
  Positive | 8 | 13 | 8 | 29
  Negative | 78 | 72 | 76 | 226

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heartburn-Free 24-Hour Periods (Day and Night) During 4 Weeks of Treatment
Description: Participants used the Reflux Symptom Questionnaire Electronic Diary (RESQ-eD) every morning upon waking and every evening before going to sleep to document the presence of daytime and nighttime heartburn and regurgitation. The percentage of heartburn-free (HBF) 24-hour periods was calculated for each participant using the following formula: (total 24-hour periods that are heartburn free / total 24-hour periods for which both a daytime and nighttime result is marked) x 100%.
Time Frame: 4 Weeks
Population: The full analysis set (FAS) included all participants randomized to a double-blind study medication. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: percentage of HBF 24-hour periods
Arm/Group | Esomeprazole 40 mg | Vonoprazan 20 mg | Vonoprazan 40 mg
Number analyzed (Participants) | 85 | 85 | 85
percentage of HBF 24-hour periods | 36.54 (35.570) | 36.69 (33.420) | 38.43 (34.793)
Statistical Analysis 1: Comparison: Esomeprazole 40 mg vs Vonoprazan 20 mg; Test type: Superiority; p = 0.7480, Wilcoxon rank-sum test — P-values were obtained using a Pearson chi-square test for each Vonoprazan treatment compared with Esomeprazole; Wilcoxon-Mann-Whitney odds estimator = 1.0584, 97.5% CI 2-sided [0.7100 to 1.5778]
Statistical Analysis 2: Comparison: Esomeprazole 40 mg vs Vonoprazan 40 mg; Test type: Superiority; p = 0.5985, Wilcoxon rank-sum test — P-values were obtained using a Pearson chi-square test for each Vonoprazan treatment compared with Esomeprazole; Wilcoxon-Mann-Whitney odds estimator = 1.0975, 97.5% CI 2-sided [0.7368 to 1.6349]

2. Secondary Outcome: Percentage of Participants With ≥1 Sustained Resolution of Heartburn During the 4-Week Treatment Period
Description: ≥1 sustained resolution of heartburn is defined as ≥7 consecutive days without both daytime and nighttime heartburn anytime during the 4-week treatment period. Daytime and nighttime heartburn were documented by all participants using the Reflux Symptom Questionnaire Electronic Diary (RESQ-eD).
Time Frame: 4 Weeks
Population: The full analysis set (FAS) included all participants randomized to a double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 40 mg | Vonoprazan 20 mg | Vonoprazan 40 mg
Number analyzed (Participants) | 86 | 85 | 85
percentage of participants | 32.6 | 30.6 | 31.8
Statistical Analysis 1: Comparison: Esomeprazole 40 mg vs Vonoprazan 20 mg; Test type: Superiority; p = 0.782, Pearson chi-square — P-values were obtained using a Pearson chi-square test for each Vonoprazan treatment compared with Esomeprazole; Miettinen-Nurminen = 0.91, 97.5% CI 2-sided [0.44 to 1.91]
Statistical Analysis 2: Comparison: Esomeprazole 40 mg vs Vonoprazan 40 mg; Test type: Superiority; p = 0.912, Pearson chi-square — P-values were obtained using a Pearson chi-square test for each Vonoprazan treatment compared with Esomeprazole; Miettinen-Nurminen = 0.96, 97.5% CI 2-sided [0.46 to 2.01]

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Description: An adverse event (AE) is any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. Reported AEs are treatment-emergent adverse events (TEAEs). A TEAE is defined as any adverse event that occurred after the first dose of study drug during the double-blind period and up to one week after completion or withdrawal from the study.
Arm/Group | Esomeprazole 40 mg | Vonoprazan 20 mg | Vonoprazan 40 mg
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/86 | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 1/86 | 0/85 | 6/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg (N=86) | Vonoprazan 20 mg (N=85) | Vonoprazan 40 mg (N=85)
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg (N=86) | Vonoprazan 20 mg (N=85) | Vonoprazan 40 mg (N=85)
Hypothyroidism (Endocrine disorders) | 0 | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
43 more participants enrolled due to lower screen failure rate in the 5 new sites and the long run in period limited predictability of enrolment in advance. Measures had been implemented maintaining scientific integrity and participant safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02743949/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02743949/SAP_001.pdf